CLINICAL TRIAL: NCT03544528
Title: Necrotic Immature Teeth Treated by Regeneration or Apexification: A 3-dimensional Analysis
Brief Title: Cone-beam Computed Tomographic (CBCT) and Regenerative Endodontic Treatment.
Acronym: Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-520-31M
Record Dates: First submitted 2018-05-04; First posted 2018-06-01 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Dental Trauma
MeSH Terms: interventions — Regeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regeneration (Experimental): This treatment aims to regenerate pulp-like tissue within the root canal space after inducing an influx of stem cells from the apical papilla that results in reestablishment of pulp protective functions.
  Interventions: Procedure: Regeneration
- Apexification (No Intervention): Traditional method. The application of Mineral Trioxide Aggregate (MTA) as an artificial apical barrier; also refer as the MTA apical plug method.

INTERVENTIONS:
Procedure: Regeneration — Apical bleeding will be induced by passing a hand instrument beyond the apical foramen to allow blood filling in the canal. Mineral trioxide aggregate will be placed directly over the coagulated blood clot.
  Arms: Regeneration

SUMMARY:
Dental trauma injuries during childhood may have an adverse impact on oral health throughout life. If trauma injuries causes pulpal necrosis, then the root stop forming. These teeth have consequently a questionable long-term survival.

Dental management of necrotic teeth with aberrant root formation represents a challenging clinical situation. The classical approach for treating these teeth includes apexification. Both apexification with Calcium hydroxide and MTA do not achieve the goals of continued root development or restoration of pulp tissue functionality.

In the last decades, a biological based approach referred as "revascularization", or "regeneration" has emerged as a biological treatment for necrotic pulps with aberrant root development. This treatment aims to regenerate pulp-like tissue within the root canal space after inducing an influx of stem cells from the apical papilla that results in reestablishment of pulp protective functions. There is evidence supporting the regeneration potential of dental tissues after regenerative endodontic treatment. However, root formation in traumatized immature teeth seems variable.

The overall goal of this study is to gain knowledge about the treatment of immature necrotic teeth in young individuals due to dental trauma. The primary goal is to compare volumetric hard tissue formation between the MTA apexification and the regeneration treatment.

DETAILED DESCRIPTION:
A randomized controlled trial, employing 34 young individuals aged 6-18 years, with immature necrotic teeth will be included. The test group will be treated by the regeneration procedure and the control group by the application of an MTA-plug. Clinical and low-dose cone-beam computed tomography scans (preoperatively and at 18-months follow-up) will be retrieved. Clinical data with information about tooth survival, absents of symptoms, resolution of infection and root development will be taken at every session.

ELIGIBILITY:
Inclusion Criteria:

* Immature teeth and confirmed pulp necrosis caused by dental trauma.
* Teeth with apical opening larger that 1mm observed in the initial CBCT.

Exclusion Criteria:

* Extensive loss of coronal tissue that require restoration with a post that will occupy the space required for blood clot formation.
* Patients who had received antibiotic treatment during the previous 3 months.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Volumetric Comparison of hard tissue formation | 18 months
  3- dimensional analysis of regenerative treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Romani Vestman, PhD, Principal Investigator — Västerbottens Läns Landsting
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No